CLINICAL TRIAL: NCT00802620
Title: Amniotic Membrane Associated With Conjunctival Autograft Versus Conjunctival Autograft for Recurrent Pterygia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Jose Alvaro Pereira Gomes, Department of Ophthalmology, Federal University of Sao Paulo (UNIFESP), Sao Paulo, Brazil.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0616/04
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Recurrent Pterygia
Keywords: Amniotic membrane; Conjunctival autograft; Recurrent pterygia; compare amniotic membrane associated with conjunctival autograft versus conjunctival autograft alone in the treatment of recurrent pterygia
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Conjunctival autograft versus conjunctival autograft treatment for recurrent pterygia — Amniotic membrane Conjunctival autograft Conjunctival autograft Recurrent pterygia

SUMMARY:
The purpose of this study is to compare amniotic membrane associated with conjunctival autograft versus conjunctival autograft alone in the treatment of recurrent pterygia.

DETAILED DESCRIPTION:
Patients with recurrent pterygia without symblepharon were randomly assigned to undertake pterygium excision followed by amniotic membrane associated with a small conjunctival autograft (2x3mm) or conjunctival autograft (approximately 5x8mm) alone. The patients were examined after 1, 7, 30, 90, 180 and 360 days after the surgery. Recurrence was considered as a fibrovascular ingrowth of 1.5 mm or more beyond the limbus with conjunctival drag.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent pterygium

Exclusion Criteria:

* Less than 15 year of age
* Symblepharon
* Glaucoma,
* Ocular Allergy
* Ocular surface disorders

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Amniotic membrane treatment for recurrent pterygia | one year